CLINICAL TRIAL: NCT01156090
Title: A Retrospective Cohort Study of Infusion Reactions Due to Vectibix
Status: Completed | Type: Observational
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: SCRI Outcomes 04
Record Dates: First submitted 2010-06-18; First posted 2010-07-02 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Infusion Reaction
Keywords: vectibix

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vectibix: patients who received at least one treatment of Vectibix

SUMMARY:
The purpose of this study is to identify approximately 100 - 150 patients who have received Vectibix (Panitumumab) in offices and clinics located in Tennessee, North Carolina, South Carolina, and North Georgia from February 2004 - April 2009. Information regarding the incidence and severity of hypersensitivity infusion reactions to Vectibix (Panitumumab)will be captured. In patients who experienced hypersensitivity reactions, the following information will also be collected: premedication, treatment cycle symptoms that were experienced during chemotherapy, changes required in subsequent Vectibix (Panitumumab) or chemotherapy treatment, and outcome of the hypersensitivity reaction.

ELIGIBILITY:
Inclusion Criteria

* All patients treated with at least one treatment of Vectibix(Panitumumab) from February 2004 -April 2009 are eligible for the study. Patients may or may not have had an infusion reaction to Vectibix (Panitumumab). Major infusion reactions are defined as rapid onset airway obstruction(bronchospasm, stridor, hoarseness), urticaria, erythema, and/or hypotension, anaphylaxis. Minor infusion reactions are defined as transient flushing or rash, urticaria, dyspnea, drug fever.
* Patients who have received treatment with an EGFR in the past are eligible.

Exclusion Criteria

* There will be no exclusions based on age, sex, medical history, or use of concomitant therapies. All charts will be abstracted for the same information, through completion of the last chemotherapy cycle.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received Vectibix (Panitumumab) in offices and clinics located in Tennessee, North Carolina, South Carolina, and North Georgia.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of Vectibix-related infusion reactions w/high rate of Erbitux-related infusion reactions | February 2004 -April 2009
  To determine the rate of Vectibix (Panitumumab)-related infusion reactions (CTCAE v3.0 grade I-IV) in geographic areas of the United States associated with a high rate of Erbitux-related infusion reactions

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Peacock, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Baptist Hospital East, Louisville, Kentucky
  - St. Louis Cancer Care, Chesterfield, Missouri
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee